CLINICAL TRIAL: NCT07193693
Title: Assessment of Barriers Limiting Optical Coherence Tomography Penetration in Actual Clinical Practice & Training (OCT2ACT) Study
Brief Title: Barriers Limiting OCT Penetration in Clinical Practice
Acronym: OCT2ACT
Status: Recruiting | Type: Observational
Sponsor: Consorzio Futuro in Ricerca (Other)
Responsible Party: Sponsor
Other Study IDs: OCT2ACT
Record Dates: First submitted 2025-09-10; First posted 2025-09-26 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Coronary Artery Disease (CAD) (E.G., Angina, Myocardial Infarction, and Atherosclerotic Heart Disease (ASHD))
Keywords: IVUS; OCT; PCI
MeSH Terms: conditions — Coronary Artery Disease; Angina Pectoris; Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cohort intracoronary imaging NO: • Inclusion criteria
  Patients undergoing clinically indicated PCI and having at least one of the following criteria (suggestive for complex PCI) without receiving intracoronary imaging:
  * Long lesion (>38 mm)
  * True bifurcation involving side-branch with a reference diameter of >2.5 mm and Medina 1.1.1
  * Left main bifurcation
    • Exclusion criteria
  * Refusal of informed consent
- Cohort intracoronary imaging YES according to guidelines recommendation: • Inclusion criteria
  Patients undergoing clinically indicated PCI with the guidance of intracoronary imaging (OCT or IVUS) and having at least one of the following criteria (suggestive for complex PCI) receiving imaging:
  * Long lesion (>38 mm)
  * True bifurcation involving side-branch with a reference diameter of >2.5 mm and Medina 1.1.1
  * Left main bifurcation
    • Exclusion criteria
  * Refusal of informed consent
- Cohort intracoronary imaging YES outside guidelines recommendation: * Inclusion criteria Patients undergoing IVUS or OCT use.
  * Exclusion criteria
    * Long lesion (>38 mm)
    * True bifurcation involving side-branch with a reference diameter of >2.5 mm and Medina 1.1.1
    * Left main bifurcation
    * Refusal of informed consent

SUMMARY:
The updated guidelines from the European Society of Cardiology (ESC) for chronic coronary syndrome (CCS) have upgraded the use of IVUS and OCT to a class IA recommendation for complex PCI, based on evidence showing a reduction in serious clinical events, including mortality, compared to conventional angiography alone. Despite this, IVUS and OCT are underutilized in daily practice due to factors such as time, cost, and limited technology availability. Investigating the reasons behind this underuse is necessary, especially now that these technologies are more accessible and cost-effective. Additionally, OCT could be particularly helpful in specific cases such as coronary bifurcations and severe calcifications, warranting further evaluation of its use in these settings.

The objective of the study OCT2ACT is to investigate:

* The main reasons/barriers limiting the use of intracoronary imaging in complex PCI cases where it is indicated as suggested by guidelines;
* The main reasons behind the selection of IVUS or OCT in such patients;
* In cases where OCT is used, how this technology can influence the procedural planning and optimization in complex clinical settings.

The participating centers will include three cohorts of patients:

1. Cohort intracoronary imaging NO: patients who meet the inclusion/exclusion criteria, but did not undergo intracoronary imaging (IVUS or OCT) due to operator's decision.

   The aim is to describe the main reasons/barriers for not using imaging.
2. Cohort intracoronary imaging YES according to guidelines recommendation: patients who meet the inclusion/exclusion criteria and underwent intracoronary imaging as recommended by guidelines.

   The aim is to understand the main reasons for the decision to use IVUS or OCT and the clinical benefits perceived by the operator.
3. Cohort intracoronary imaging YES outside guidelines recommendation: patients who meet the inclusion/exclusion criteria and underwent intracoronary imaging (IVUS or OCT) outside.

DETAILED DESCRIPTION:
The last update of European Society of Cardiology (ESC) chronic coronary syndrome (CCS) guidelines upgraded the use of intravascular ultrasound (IVUS) imaging and optical coherence tomography (OCT) to class IA in the setting of complex percutaneous coronary intervention (PCI) (in particular left main, true bifurcations, and long lesions).

This strong level of recommendation is based on the recent evidence that intracoronary imaging reduces the incidence of hard clinical endpoints, including mortality, as compared to conventional angiography alone.

Yet, there is compelling evidence documenting the under-utilization of IVUS and OCT in daily practice. Many potential reasons, including time, costs, limited availability of technology, expertise of the operators have been suggested. However, no specific study investigated the reasons behind this malpractice. In particular, these reasons should be investigated now that intracoronary imaging has been upgraded to class I recommendation and that many technologies are available significantly reducing the economic burden. In addition, there are some particular anatomic subsets where OCT could be particularly helpful (bifurcations, severe calcification, acute coronary syndrome patients) and it could be interesting to assess the penetration of this technology in this subset of patients. Finally, these devices can be used also in anatomical subsets (diagnosis and procedural guidance) outside from Guidelines recommendations and it is important to assess their safety and clinical advantage in this setting.

Objective

The OCT2ACT study aims to investigate:

* The main reasons/barriers limiting the use of intracoronary imaging in complex PCI where it is indicated as suggested by guidelines
* The main reasons behind the selection of IVUS or OCT in complex PCI
* In complex PCI guided by OCT, How OCT can influence the procedural planning and optimization in complex clinical settings.

The OCT2ACT is an observational, prospective, multicenter, investigator-driven study.

Participating centers will include three different cohorts of patients:

1. Cohort intracoronary imaging NO In this cohort, the investigators will include all the patients matching inclusion/exclusion criteria, but in whom intracoronary imaging (IVUS or OCT) was not used (operator's decision). The aim is to have a description of the main reasons/barriers that led to the avoidance of imaging utilization.
2. Cohort intracoronary imaging YES according to guidelines recommendation In this cohort, the investigators will include all the patients matching inclusion/exclusion criteria in whom intracoronary imaging (IVUS or OCT) was used (operator's decision) according to guidelines recommendation. The aim is to understand the main reasons behind the decision to use IVUS or OCT and the clinical advantages perceived by the operators.
3. Cohort intracoronary imaging YES outside guidelines recommendation In this cohort, the investigators will include all the patients matching inclusion/exclusion criteria in whom OCT was used (operator's decision) outside Guidelines recommendations. The aim is to understand the main reasons behind the decision to use OCT outside guidelines recommendation, its safety and the clinical advantages perceived by the operators.

After Ethic Committee approval and site initiation visit, each participating center will recruit consecutive patients for a time window of 3 months.

ELIGIBILITY:
1. Cohort intracoronary imaging NO

   • Inclusion criteria

   Patients undergoing clinically indicated PCI and having at least one of the following criteria (suggestive for complex PCI) without receiving intracoronary imaging:
   * Long lesion (>38 mm)
   * True bifurcation involving side-branch with a reference diameter of >2.5 mm and Medina 1.1.1
   * Left main bifurcation

     • Exclusion criteria
   * Refusal of informed consent
2. Cohort intracoronary imaging YES according to guidelines recommendation

   • Inclusion criteria

   Patients undergoing clinically indicated PCI with the guidance of intracoronary imaging (OCT or IVUS) and having at least one of the following criteria (suggestive for complex PCI) receiving imaging:
   * Long lesion (>38 mm)
   * True bifurcation involving side-branch with a reference diameter of >2.5 mm and Medina 1.1.1
   * Left main bifurcation

     • Exclusion criteria
   * Refusal of informed consent
3. Cohort intracoronary imaging YES outside guidelines recommendation

   * Inclusion criteria Patients undergoing IVUS or OCT use.
   * Exclusion criteria

     * Long lesion (>38 mm)
     * True bifurcation involving side-branch with a reference diameter of >2.5 mm and Medina 1.1.1
     * Left main bifurcation
     * Refusal of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing PCI and receiving or not receiving imaging according to ESC indication guidelines. Patients undergoing coronary artery angiography and/or PCI and receiving imaging in a setting outside from ESC indication guidelines.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2025-12-15 (Actual); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
Cohort intracoronary imaging NO: Reasons/barriers for not using intracoronary imaging | From the enrollment to the end of the procedure
  As suggested in the consensus document by Cabana et al, the main reasons/barriers will be classified according to the following groups:
  Attitudes (lack of agreement and inertia of previous practice):
  * Clinical and angiographic data are sufficient
  * Intracoronary imaging would not change my PCI strategy
  * Intracoronary imaging has low added value on improving clinical outcome
  Knowledge (lack of awareness and familiarity):
  * Intracoronary imaging not feasible for technical or anatomical reasons (e.g., tortuous vessels, etc.)
  * Lack of confidence in interpretation of images
  * Lack of confidence in translating imaging features into an actionable PCI plan
  * Inadequate support by device specialists in the cath lab
  Behavior (external barriers):
  * Time constraint
  * Device costs
  * Absence of adequate coding / reimbursement
Cohort intracoronary imaging YES according to guidelines recommendations: Reasons behind the selection of IVUS or OCT | From enrollment to the end of the procedure
  The operator has to define the reason behind the choice of the imaging modality with particular regard to the anticipated benefit related to such choice.
Cohort intracoronary imaging YES outside guidelines recommendations: Reasons behind the selection of OCT or IVUS outside guidelines recommendations | from enrollment to the end of the procedure
  The operator has to define the reason behind the choice of the imaging modality with particular regard to the anticipated benefit related to such choice in a setting that is outside guidelines recommendations

SECONDARY OUTCOMES:
Cohort intracoronary imaging NO: secondary endpoints | from September to December 2025
  Percentage of PCI matching inclusion/exclusion criteria
Cohort intracoronary imaging NO: secondary endpoints | from September to December 2025
  Percentage of PCI where intracoronary imaging is used as compared to overall volume of PCI
Cohort intracoronary imaging NO: secondary endpoints | from September to December 2025
  Percentage of PCI where intracoronary imaging is used as compared to overall volume of PCI matching inclusion/exclusion criteria
Cohort intracoronary imaging NO: secondary endpoints | from September to December 2025
  Association between baseline and procedural characteristics and missing use of intracoronary imaging
Cohort intracoronary imaging YES outside guidelines recommendations: safety endpoints | from enrollment to the end of the procedure
  Procedural time. The safety endpoints will be recorded in both the cohorts intracoronary imaging YES and compared to investigate differences.
Cohort intracoronary imaging YES outside guidelines recommendations: safety endpoints | from enrollment to the end of the procedure
  Contrast media amount. The safety endpoints will be recorded in both the cohorts intracoronary imaging YES and compared to investigate differences.
Cohort intracoronary imaging YES outside guidelines recommendations: safety endpoints | from enrollment to the end of the procedure
  Procedural complications related to OCT or IVUS use. The safety endpoints will be recorded in both the cohorts intracoronary imaging YES and compared to investigate differences.
Cohort intracoronary imaging YES outside guidelines recommendations: secondary endpoints | from September to December 2025
  Association between baseline and procedural characteristics and IVUS/OCT preference
Cohort intracoronary imaging YES outside guidelines recommendations: secondary endpoints | from September to December 2025
  Description of timing and modality of the intracoronary imaging
Cohort intracoronary imaging YES outside guidelines recommendations: secondary endpoints | from September to December 2025
  Description of the operator's perceived advantages by intracoronary imaging use
Cohort intracoronary imaging YES outside guidelines recommendations: secondary endpoints | from September to December 2025
  Description of OCT penetration over IVUS in bifurcations, LM and stent failure

CONTACTS AND LOCATIONS:
Overall Officials: Simone Biscaglia, Study Chair — Azienda Ospedaliero Universitaria di Ferrara; Vergallo Rocco, Principal Investigator — Ospedale Policlinico San Martino; Paolo Canova, Principal Investigator — ASST Papa Giovanni XXIII, Bergamo
Locations (2):
- Italy (2):
  - ASST Papa Giovanni XXIII, Bergamo
  - Ospedale San Martino, Genova

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vrints C, Andreotti F, Koskinas KC, Rossello X, Adamo M, Ainslie J, Banning AP, Budaj A, Buechel RR, Chiariello GA, Chieffo A, Christodorescu RM, Deaton C, Doenst T, Jones HW, Kunadian V, Mehilli J, Milojevic M, Piek JJ, Pugliese F, Rubboli A, Semb AG, Senior R, Ten Berg JM, Van Belle E, Van Craenenbroeck EM, Vidal-Perez R, Winther S; ESC Scientific Document Group. 2024 ESC Guidelines for the management of chronic coronary syndromes. Eur Heart J. 2024 Sep 29;45(36):3415-3537. doi: 10.1093/eurheartj/ehae177. No abstract available. PMID 39210710